CLINICAL TRIAL: NCT05750615
Title: Understanding Factors Which Affect Willingness to Self-manage a Pessary for Pelvic Organ Prolapse: A Mixed Methods Study Aiming to Improve Access to Pessary Self-management.
Brief Title: What Affects Willingness to Self-manage a Pessary?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B01328
Record Dates: First submitted 2022-08-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Prolapse; Female; Prolapse, Vaginal
MeSH Terms: conditions — Prolapse; Uterine Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Quantitative phase: Pessary using women
- Qualitative phase: Pessary using women
- Intervention development phase: Pessary using women and pessary practitioners
- Pilot phase: Pessary using women
  Interventions: Other: Uncertain what intervention will be co-created

INTERVENTIONS:
Other: Uncertain what intervention will be co-created — Uncertain what intervention will be co-created
  Groups: Pilot phase

SUMMARY:
Pessary self-management is defined as the patient's ability to remove and reinsert their pessary themselves at home. Previous research has suggested that some women may prefer being able to remove and reinsert their pessary as they wish rather than wait for clinic appointments. At the moment, not enough is known about pessary self-management, particularly what makes someone more or less likely to try pessary self-management. The investigators would like to understand this better to try to help women overcome barriers they might face. This study aims to collect data via both questionnaires and interviews to explore willingness to self-manage a pessary. Using findings from the questionnaires and interviews, a group of women who use pessaries and healthcare professionals who provide pessary care will work together to develop a better way to support women to feel able and willing to manage their pessary in future.

ELIGIBILITY:
Quantitative phase inclusion criteria

* Willing and able to give implied consent by completion of the questionnaire
* Female
* Over the age of 18 years
* Have retained a pessary for pelvic organ prolapse for a minimum of two weeks
* Able to speak and understand English
* Use a ring, shaatz, cube or inflatable pessary

Qualitative phase inclusion criteria

* Willing and able to give informed consent
* Female
* Over the age of 18 years
* Have retained a pessary for pelvic organ prolapse for a minimum of two weeks
* Speak English or, for those whose first or preferred language is a language other than English, speak a language there is an available interpreter for

Intervention development phase inclusion criteria Pessary using women

* Willing and able to give informed consent
* Female
* Over the age of 18 years
* Have retained a pessary for pelvic organ prolapse for a minimum of two weeks
* Speak English Pessary practitioners
* Willing and able to give informed consent
* Provide regular pessary care as part of clinical role (defined as insertion or removal of a woman's pessary on a minimum of a monthly basis)
* Speak English

Pilot phase inclusion criteria

* Willing and able to give informed consent, review the intervention and provide written and/or verbal feedback.
* Female
* Over the age of 18 years
* Have retained a pessary for pelvic organ prolapse for a minimum of two weeks
* Speak English
* Have no previous experience self-managing a pessary (defined as never having removed or inserted their pessary, or received any pessary self-management teaching or support from a healthcare professional)

Exclusion Criteria:

Quantitative phase exclusion criteria

* Lacking capacity to give implied consent by completion of the questionnaire
* Has a first or preferred language that is not English
* Use a shelf, gell-horn or donut pessary

Qualitative phase exclusion criteria

* Lacking capacity to give informed consent
* First or preferred language that is not English or a language there is an available interpreter for

Intervention development phase exclusion criteria Pessary using women

* Lacking capacity to give informed consent
* Does not speak English Pessary practitioners
* Lacking capacity to give informed consent
* Does not speak English
* Does not provide pessary care at a minimum of a monthly basis

Intervention pilot exclusion criteria

* Lacking capacity to give informed consent, review the intervention and provide written and/or verbal feedback.
* Does not speak English
* Have prior experience self-managing a pessary (defined as previously removing or inserting their pessary, or receiving any pessary self-management teaching or support from a healthcare professional)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pessary using women and pessary practitioners
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Willingness to self-manage a pessary | Through study completion, an average of 1 appointment (1 day)
  Women will be asked whether they are willing or not to self-manage a pessary for prolapse. This will be a binary yes, no or not sure answer.

SECONDARY OUTCOMES:
Age | Through study completion, an average of 1 appointment (1 day)
  Full years since birth
Pessary | Through study completion, an average of 1 appointment (1 day)
  Type and size of pessary in situ
Length of pessary management | Through study completion, an average of 1 appointment (1 day)
  Total months pessary used for
Comorbidities | Through study completion, an average of 1 appointment (1 day)
  Free text data for participant to report diagnosed health conditionns
Self-management experience | Through study completion, an average of 1 appointment (1 day)
  The woman will be asked whether she has previously removed or inserted her pessary
Self-management status | Through study completion, an average of 1 appointment (1 day)
  The woman will be asked whether she is currently self-managing her pessary (defined as removing and inserting it independently in between clinic appointments)
Ethnicity | Through study completion, an average of 1 appointment (1 day)
  Ethnic groups in accordance with UK government agreed list of ethnicities
Post code | Through study completion, an average of 1 appointment (1 day)
  Post code at home address to determine deprivation of home address in accordance with UK government index of deprivation
Education status | Through study completion, an average of 1 appointment (1 day)
  Women will be asked to report their highest level of education
Female genital self-image score (FGSIS) | Through study completion, an average of 1 appointment (1 day)
  Women will also be asked to complete the Female Genital Self-Image Scale (FGSIS-4), a reliable and validated 4-item questionnaire which measures women's attitude and beliefs about their genitals (Herbenick and Reece, 2010). Scores in the FGSIS-4 range between 4-16, with a mean score of 12 in a nationally representative population of over 2000 American women (Herbenick et al., 2011). Herbenick et al. (2011) have not determined a binary score for high and low FGSIS, however for the purpose of this study, a score of eight or less will indicate low FGSI, whereas more than eight will indicate high FGSI. To score eight or less, a participant must disagree with all four statements describing genital self-image therefore this is deemed to accurately represent FGSIS-4.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT05750615/Prot_SAP_000.pdf